CLINICAL TRIAL: NCT02067819
Title: Proof of Concept Study of an Oral Orthotic to Reduce Tic Severity in Chronic Tic Disorder and Tourette Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: The Hindin Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1208012905
Record Dates: First submitted 2014-02-18; First posted 2014-02-20 (Estimated); Results first posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-04

CONDITIONS: Tourette Syndrome; Chronic Tic Disorder
Keywords: Tourette's; Tic Disorder; Dental Appliance; Oral Orthotic; Mouthguard
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders | interventions — Occlusal Splints; Orthotic Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active Oral Orthotic Treatment (Experimental): Active treatment group will receive an occlusal splint adjusted to the appropriate therapeutic height (based on an initial fitting). Participants will be instructed to wear the orthotic 24/7 (or as close as possible) for the duration of the study.
  Interventions: Device: Active Oral Orthotic Treatment
- Placebo Oral Orthotic Treatment (Placebo Comparator): Control participants will receive an identical sham splint to the active condition, but not adjusted to the recommended height for the given participant. Participants will be asked to wear the orthotic 24/7 for the duration of the study.
  Interventions: Device: Placebo Oral Orthotic Treatment

INTERVENTIONS:
Device: Active Oral Orthotic Treatment — Active treatment group will receive an occlusal splint adjusted to the appropriate therapeutic height (based on an initial fitting). Participants will be instructed to wear the orthotic 24/7 (or as close as possible) for the duration of the study.
  Other Names: Occlusal Splint; Oral Orthotic; Dental Orthotic; Dental Appliance
  Arms: Active Oral Orthotic Treatment
Device: Placebo Oral Orthotic Treatment — After two weeks, this treatment group will receive an occlusal splint adjusted to the appropriate therapeutic height (based on an initial fitting). Participants will be instructed to wear the orthotic 24/7 (or as close as possible) for the duration of the study.
  Arms: Placebo Oral Orthotic Treatment

SUMMARY:
The purpose of this study is to assess the feasibility of a trial on an oral orthotic for reducing tic severity in children ages 7-25 years with Tourette syndrome (TS) or Chronic Tic Disorder (CTD).

DETAILED DESCRIPTION:
The study is a 2 group, 2 week randomized controlled feasibility trial of an active vs sham oral orthotic to reduce tic severity in children and adolescents ages 7-25 years. Responders to acute phase treatment will be followed for 10 additional week (12 weeks total) to assess intervention durability, safety and acceptability. Non-responders to the sham orthotic will be provided active treatment at the end of the 2 week acute phase. We aim to assess and enroll 24 participants; twelve participants will receive an orthotic adjusted to the appropriate therapeutic height, and twelve participants will receive an identical sham orthotic, but not adjusted to the recommended height for the given participant.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-25 inclusive.
* Presence of motor and/or vocal tics for at least 12 months.
* Tics are of at least moderate clinical severity as evidenced by a Yale Global Tic Severity score of 14 or higher for motor or vocal tics only and 22 or higher for Tourette syndrome and present during the baseline assessment.
* IQ estimate of 70 or higher
* Comorbid disorder (e.g., ADHD, OCD, ODD) will be allowed provided that the tic symptoms are of primary concern to parents and comorbid symptoms are not of sufficient severity to require immediate treatment other than that provided by the current study.
* Pre-existing stable medication (see protocol for details), tic or otherwise, will also be allowed provided the family agrees to refrain from med changes over the course of the acute phase of the study
* Sufficient command of the English language to participate in informed consent and assessment procedures.
* Agree for videotaping of study procedures
* Clearance by treating dentist: Certification of good dental health provided by the subjects current dentist prior to enrollment in the study

Exclusion Criteria:

* Major psychiatric disorder at screening that would preclude full participation in study procedures including psychosis, mania, depression, untreated combined type ADHD, autism and pervasive developmental disorders.
* Medication changes are planned during the acute and follow-up phase of treatment.
* Other dental health problems that might interfere with the assessment, installation, or wearing of orthotic device.
* Does not consent to being videotaped

Ages: 7 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2014-03; Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Bennett, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Oral Orthotic Treatment | Placebo Oral Orthotic Treatment
Started | 11 | 10
Completed | 6 | 7
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Oral Orthotic Treatment | Placebo Oral Orthotic Treatment | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.27 (5.293) | 12.5 (4.90) | 12.38 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Global Severity of Tics and Clinical Condition as Measured by YGTSS
Description: The primary clinical outcome measures included the Yale Global Tic Severity Scale (YGTSS). The YGTSS is a semi structured interview designed to elicit information regarding the character & anatomical distribution of tics observed during the course of 1 week interval, prior to clinical assessment. Following completion of the interview & construction of a "tic inventory", clinicians rate severity of motor and photic tics along with 5 separate dimensions (frequency, intensity, number, complexity, interference).
  The YGTSS is comprised of a list of motor and vocal tics & the participant endorses which tics are currently present. Motor and vocal tics are then separately rated for Number, Frequency, Intensity, Complexity, Interference & Impairment, each on a 6 point likert scale ranging from 0 (none) to 5 (Severe).This results in a range of 0-25 for motor tics & 0-25 for vocal tics, for a total score range of 0-50. A score of 0 indicating a lack of tics & 50 represent the most severe tics.
Time Frame: Baseline Visit, Week 2 Visit
Population: 4 opted not to participate after randomization but prior to receiving the orthotic. 1 participant dropped out after baseline visit due to belief that oral orthotic was responsible for disruptive behavior at school. 1 participant was removed from study at Baseline by PI due to medication change for bipolar d/o. 1 participant dropped out after Week 2 due to discomfort when wearing the oral orthotic.1 patient failed to respond to attempted contact from the study team following baseline visit
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Oral Orthotic Treatment | Placebo Oral Orthotic Treatment
Number analyzed (Participants) | 6 | 7
score on a scale | 20.19 (1.06) | 25.82 (0.99)

2. Secondary Outcome: Change in Number, Frequency, and Intensity of Motor and Vocal Tics as Measured by the Clinical Global Impressions Scale - Severity
Description: To assess global severity of tics and change in the clinical condition over time, the Clinical Global Impressions Scale - Severity (CGI-S) was utilized. The Severity of Illness has a low score of 0 and high score is 7. The low score of 0 represents that the subject was not assessed and the high score of 7 represents among the most extremely ill subjects.
Time Frame: Baseline Visit, Week 2 Visit
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Oral Orthotic Treatment | Placebo Oral Orthotic Treatment
Number analyzed (Participants) | 6 | 7
score on a scale | 4.57 (0.25) | 5.27 (0.23)

ADVERSE EVENTS:
Time Frame: Ten Weeks
Description: Participants reported all side effects or adverse events in a diary at home, as well as on a structured adverse events questionnaire during study visits. Study personnel additionally inquired about adverse events at each visit. The total number of participants at risk for an adverse event was 17, because 17 participants received the oral orthotic (8 were active, 9 were placebo).
Arm/Group | Active Oral Orthotic Treatment | Placebo Oral Orthotic Treatment
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 6/8 | 6/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Oral Orthotic Treatment (N=8) | Placebo Oral Orthotic Treatment (N=9)
mouth soreness (Social circumstances) | 6 (6) | 6 (6) — mild to moderate jaw pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT02067819/Prot_000.pdf